CLINICAL TRIAL: NCT05032638
Title: Promoting Adherence in Upper Extremity Home-based Rehabilitation Through Motivational Interviewing and Ecological Momentary Assessment
Brief Title: Adherence in Upper Extremity Home-based Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-00513
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Stroke
Keywords: Stroke; upper extremity; motivational interviewing; shared decision making; ecological momentary assessments; self-initiated training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Subjects with motor impairment will work closely with an occupational therapist to identify a goal and select activities that they will work on at home to improve the function of their affected arm.
  Interventions: Behavioral: Therapist guided training; Behavioral: Upper extremity (UE) Training

INTERVENTIONS:
Behavioral: Therapist guided training — Therapist guided period delivered virtually (WebEx/Zoom). Participants will be patients associated with NYULH and will have access to Zoom. Each session will last 45 min, and will completed 3x/week by research therapists, who are part of the study.
Behavioral: Upper extremity (UE) Training — The 4-week UE training is completed in the participants home on their own and communication with study staff is virtual. Participants will receive daily communication through the Expiwell app to answer survey questions related to adherence, and safety/adverse events. Participants will also complete weekly check-ins with their research therapist over Zoom to answer questions about difficulties related to UE training activities, refinement of training goals, and to receive feedback on their training performance. Each weekly check-in will be approximately 45 minutes.

SUMMARY:
The objective of the proposal is to determine the feasibility of implementing Ecological Momentary Assessment (EMA) and Motivational Interviewing (MI) methods to enhance adherence for a 4-week self-initiated arm training protocol. A non-randomized feasibility study using a 4-week UE training protocol will be conducted in 15 individuals within the first 12 months post-stroke living in the community. EMA data will be collected using a mobile app to automate real-time collection of adherence data on a daily basis. MI will be used to produce self-generated training plans (training goals, training schedule), guided by the therapist before the start of training.

DETAILED DESCRIPTION:
Using a mixed methods design, the study will collect quantitative data before, during, and after training. Qualitative data will be collected after the training period and analyzed to explain the quantitative findings in depth, within the context of everyday life. Study aim 1 is to evaluate the feasibility of using EMA to measure adherence and of applying the MI approach. Quantitative data will include four indicators of adherence and accuracy. Interview responses will be used as qualitative data to elucidate participants' acceptance of the MI approach and feedback on using the EMA app. Study aim 2 is to explore to what extent UE outcomes change after the 4-week self-initiated home-based rehabilitation program. Outcomes will include UE use in real-world environments and self-perceived changes in UE use.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years old) diagnosed with stroke at least 6 months ago at the time of screening
* Living in the community
* Have presence of UE motor impairment on the affected side (Fugl-Meyer Assessment scores < 66)
* Availability of mobile technology (tablet or smartphone) with internet connection to use phone app and Zoom videochat)
* Be medically stable
* Able to provide written consent

Exclusion Criteria:

* Currently receiving active occupational or physical therapy for the treatment of the affected UE
* Presence of severe cognitive impairment (Mini Mental Status Exam <24)
* Self-reported moderate to severe pain of the affected UE with use
* Presence of unilateral spatial neglect (Star Cancellation Task scores < 44)
* Presence of neurological diagnosis other than stroke.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Rates of adherence at individual and group level measured through frequency | Day 4 visit
  Frequency will be calculated by dividing the number of sessions completed by the total number of sessions available for 4-week period
Rates of adherence at individual and group level measured through frequency | Day 6 visit
  Frequency will be calculated by dividing the number of sessions completed by the total number of sessions available for 4-week period
Rates of adherence at individual and group level measured through frequency | Day 8 visit
  Frequency will be calculated by dividing the number of sessions completed by the total number of sessions available for 4-week period
Rates of adherence at individual and group level measured through frequency | Day 11 visit
  Frequency will be calculated by dividing the number of sessions completed by the total number of sessions available for 4-week period
Rates of adherence at individual and group level measured through frequency | Day 22 visit
  Frequency will be calculated by dividing the number of sessions completed by the total number of sessions available for 4-week period
Rates of adherence at individual and group level measured through frequency | Day 29 visit
  Frequency will be calculated by dividing the number of sessions completed by the total number of sessions available for 4-week period
Rates of adherence at individual and group level measured through frequency | Day 37 visit
  Frequency will be calculated by dividing the number of sessions completed by the total number of sessions available for 4-week period
Rates of adherence at individual and group level measured through frequency | Day 39 visit
  Frequency will be calculated by dividing the number of sessions completed by the total number of sessions available for 4-week period
Rates of adherence at individual and group level measured through intensity | Day 4 visit
  Intensity data will be collected using a 3-point ordinal ratings scale to determine perceived intensity of practice for each session (mild- moderate- intense).
Rates of adherence at individual and group level measured through intensity | Day 6 visit
  Intensity data will be collected using a 3-point ordinal ratings scale to determine perceived intensity of practice for each session (mild- moderate- intense).
Rates of adherence at individual and group level measured through intensity | Day 8 visit
  Intensity data will be collected using a 3-point ordinal ratings scale to determine perceived intensity of practice for each session (mild- moderate- intense).
Rates of adherence at individual and group level measured through intensity | Day 11 visit
  Intensity data will be collected using a 3-point ordinal ratings scale to determine perceived intensity of practice for each session (mild- moderate- intense).
Rates of adherence at individual and group level measured through intensity | Day 22 visit
  Intensity data will be collected using a 3-point ordinal ratings scale to determine perceived intensity of practice for each session (mild- moderate- intense).
Rates of adherence at individual and group level measured through intensity | Day 29 visit
  Intensity data will be collected using a 3-point ordinal ratings scale to determine perceived intensity of practice for each session (mild- moderate- intense).
Rates of adherence at individual and group level measured through intensity | Day 37 visit
  Intensity data will be collected using a 3-point ordinal ratings scale to determine perceived intensity of practice for each session (mild- moderate- intense).
Rates of adherence at individual and group level measured through intensity | Day 39 visit
  Intensity data will be collected using a 3-point ordinal ratings scale to determine perceived intensity of practice for each session (mild- moderate- intense).
Rates of adherence at individual and group level measured through duration | Day 4 visit
  Duration data will be collected using open end responses to report total number of minutes of UE training completed that day
Rates of adherence at individual and group level measured through duration | Day 6 visit
  Duration data will be collected using open end responses to report total number of minutes of UE training completed that day
Rates of adherence at individual and group level measured through duration | Day 8 visit
  Duration data will be collected using open end responses to report total number of minutes of UE training completed that day
Rates of adherence at individual and group level measured through duration | Day 11 visit
  Duration data will be collected using open end responses to report total number of minutes of UE training completed that day
Rates of adherence at individual and group level measured through duration | Day 22 visit
  Duration data will be collected using open end responses to report total number of minutes of UE training completed that day
Rates of adherence at individual and group level measured through duration | Day 29 visit
  Duration data will be collected using open end responses to report total number of minutes of UE training completed that day
Rates of adherence at individual and group level measured through duration | Day 37 visit
  Duration data will be collected using open end responses to report total number of minutes of UE training completed that day
Rates of adherence at individual and group level measured through duration | Day 39 visit
  Duration data will be collected using open end responses to report total number of minutes of UE training completed that day
Decision making factors effecting the program adherence through semi-structured interviews | Day 39 visit
  Semi-structured interviews will be conducted with all participants to collect qualitative data on participants' experiences related to the shared decision-making process in phase 1, and adherence to arm training in phase 2 of study.

SECONDARY OUTCOMES:
Change scores in Fugl-Meyer Assessment from baseline to discharge and baseline to follow-up | Day 4 visit, Day 37-39 visit, Day 65-67 visit
  FMA is a valid and reliable UE assessment to measure motor impairment in stroke. It consists of 33 items reflecting typical shoulder and hand motions in and out of synergy patterns characteristic of motor recovery after stroke. It is the gold standard performance-based assessment in UE stroke rehabilitation with an established minimal clinically important difference (MCID) of 4.25-7.25 points for chronic stroke patients.
Change scores in Motor Activity Log from baseline to discharge and baseline to follow-up | Day 4 visit, Day 37-39 visit, Day 65-67 visit
  Motor Activity Log (MAL) is a valid and reliable self-report questionnaire for individuals in the subacute and chronic phase after stroke. Originally created as the primary outcome for Constraint Induced Movement Therapy, the MAL captures spontaneous use of the affected UE in daily life. It consists of 28 items reflecting basic and instrumental activities of daily living items. Scoring is based on an ordinal scale ranging from 1-5, and final scores are determined by calculating the mean of all item scores. This study will use the amount of use subscale for this study.
Change scores in Canadian Occupational Performance Measure from baseline to discharge and baseline to follow-up | Day 4 visit, Day 37-39 visit, Day 65-67 visit
  The Canadian Occupational Performance Measure (COPM) is a valid and reliable individualized self-report measure that quantifies a participants' perception of everyday performance. Participants rate their change in their performance and satisfaction on a scale of 1 (unable to perform/not satisfied) to 10 (able to perform, extremely satisfied). A change of two or more points is considered clinically significant.
Change scores in UE accelerometry data calculated using bilateral magnitude ratio from baseline to discharge and baseline to follow-up. | Day 4 visit, Day 37-39 visit, Day 65-67 visit
  Wrist worn accelerometers can be used to provide objective, valid, and reliable data on general UE motion in home settings. As a secondary outcome for adherence, we will collect bilateral UE accelerometry data continuously for 24 hours at all timepoints to determine if there are any changes in UE motion of the affected side in relation to the unaffected side before and after the intervention. Commercially available Actigraph GT9X Link wrist sensors will be used to collect bilateral UE motion at baseline, discharge, and follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Kim, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.The investigator who proposed to use the data.
Access Criteria: Upon reasonable request. Requests should be directed to gjk207@nyu.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Kim GJ, Gahlot A, Magsombol C, Waskiewicz M, Capasso N, Van Lew S, Goverover Y, Dickson VV. Protocol for a remote home-based upper extremity self-training program for community-dwelling individuals after stroke. Contemp Clin Trials Commun. 2023 Mar 17;33:101112. doi: 10.1016/j.conctc.2023.101112. eCollection 2023 Jun. PMID 37113325